CLINICAL TRIAL: NCT00135460
Title: Comparing a Nucleoside-Analogue-Sparing Regimen and a Protease-Inhibitor-Sparing Regimen in Patients With HIV. Influence on Morphological and Metabolic Disorders. A Randomized, Open-Label Multicenter Trial.
Brief Title: Comparing a Nucleoside-Analogue-Sparing Regimen and a Protease-Inhibitor-Sparing Regimen in HIV Infected Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish HIV Research Group (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2612-2198
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2005-09

CONDITIONS: HIV-Associated Lipodystrophy Syndrome
Keywords: HIV; Lipoatrophy; Lipodystrophy; Treatment Naive; HIV Infections; Hypercholesterolemia
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Lipodystrophy; HIV Infections; Hypercholesterolemia

INTERVENTIONS:
Drug: nucleoside analogue sparing HAART regimen

SUMMARY:
Highly active antiretroviral therapy (HAART) has improved the long time survival of HIV infected individuals. However an increasing number of HIV-patients have developed metabolic and morphological alterations including peripheral lipoatrophy.

There is limited knowledge about lipodystrophic adverse events in nucleoside reverse transcriptase inhibitor (NRTI)-sparing regimens. The hypothesis is that nucleoside analogues are responsible for development of lipoatrophy, and, patients receiving an NRTI-sparing regimen will have little risk of peripheral lipoatrophy.

The researchers plan to perform a randomized study recruiting 100 antiretroviral naive patients that will be randomized to receive a nucleoside analogue sparing HAART regimen or a protease-inhibitor sparing regimen.

The main endpoint is changes in peripheral fat mass as determined by dual energy X-ray absortiometry (DEXA)-scanning.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral naïve patients
* HIV-1 infection as documented by a licensed HIV-1 antibody ELISA.
* Fulfilling the criteria for starting antiretroviral therapy.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Women being pregnant or breast-feeding.
* Fertile women using no safe contraception.
* Patients with active intravenous drug use.
* Abuse of alcohol, which in the opinion of the treating physician will reduce the patient´s ability to follow a therapeutic regimen and evaluations of the protocol.
* Ongoing medical treatment, which has a clinically significant interaction with lopinavir, ritonavir or efavirenz.
* Creatinine > 200 mmol/l.
* ALT or AST > 5 times upper normal value (200U/l).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-06; Study Completion 2007-11

PRIMARY OUTCOMES:
Changes in peripheral fat mass, determined by DEXA-changes
Changes in body composition from baseline, determined by patient and physician in a standardized questionnaire and by standardized clinical examination
Change from baseline in fasting lipids and subsets hereof
Development of impaired glucose tolerance and insulin resistance

SECONDARY OUTCOMES:
Proportion of patients with HIV-RNA < 20 copies after 24, 48, 72 and 96 weeks
Change in CD4 cell count from baseline after 24, 48, 72 and 96 weeks
Incidence of adverse events
Incidence of clinical disease progression
Proportion of patients who have virological, immunological or clinical failure or treatment-limiting adverse events at week 24, 48 and 96
Change in plasma lactate from baseline
Time to discontinuation of the randomized therapy and reasons for this
Incidence of genotypical and virological resistance
Development of osteopenia, judged by DEXA-scan
Compliance - proportion of patients who report to take 90%, respectively 95% of their medications at week 4, 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gerstoft, M.D., DMSc, Study Chair — Rigshospitalet, Denmark; Niels Obel, M.D., DMSc, Principal Investigator — Odense University Hospital; Court Pedersen, Professor, Principal Investigator — Odense University Hospital; Lars Mathiesen, M.D.,DMSc, Principal Investigator — Hvidovre University Hospital; Henrik Nielsen, M.D.,DMSc, Principal Investigator — Aalborg University Hospital; Alex Laursen, M.D., DMSc, Principal Investigator — Aarhus University City; Ann-Brit E Hansen, M.D., Principal Investigator — Copenhagen University Hospital Rigshospitalet and Odense University Hospital
Locations (5):
- Denmark (5):
  - Department of Infectious Diseases, Hvidovre University Hospital, Hvidovre, Copenhagen
  - Department of Infectious Diseases, Aalborg Hospital, Aalborg
  - Department of Infectious Diseases, Aarhus University Hospital, Aarhus
  - Department of Infectious Diseases, Rigshospitalet, Copenhagen
  - Department of Infectious Diseases, Odense University Hospital, Odense

REFERENCES:
- [Derived] Mathiesen IH, Salem M, Gerstoft J, Gaardbo JC, Obel N, Pedersen C, Ullum H, Nielsen SD, Hansen AE. Complete manuscript Title: Changes in RANKL during the first two years after cART initiation in HIV-infected cART naive adults. BMC Infect Dis. 2017 Apr 11;17(1):262. doi: 10.1186/s12879-017-2368-y. PMID 28399815